CLINICAL TRIAL: NCT01822613
Title: A Phase Ib/II, Open-label Study of LJM716 in Combination With BYL719 Compared to Taxane or Irinotecan in Patients With Previously Treated Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Study of Safety & Efficacy of the Combination of LJM716 & BYL719 in Patients With Previously Treated Esophageal Squamous Cell Carcinoma (ESCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLJM716X2103
Record Dates: First submitted 2013-03-22; First posted 2013-04-02 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — elgemtumab; Alpelisib; Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LJM716-BYL719 arm (Experimental): approximately 42 previously treated esophageal squamous cell carcinoma (ESCC) patients will be enrolled to the LJM716-BYL719 combination arm to evaluate the anti-tumor activity and further assess the safety, tolerability and anti-tumor activity of the combination versus current therapies (physician's choice of paclitaxel, docetaxel or irinotecan).
  Interventions: Drug: LJM716; Drug: BYL719
- Paclitaxel, Docetaxel or Irinotecan arm (Active Comparator): approximately 42 previously treated esophageal squamous cell carcinoma (ESCC) patients will be enrolled to the Paclitaxel, Docetaxel or Irinotecan arm (physician's choice arm) to evaluate the anti-tumor activity and further assess the safety, tolerability and anti-tumor activity of the LJM716-BYL719 combination versus current therapies (physician's choice of paclitaxel, docetaxel or irinotecan).
  Interventions: Drug: Paclitaxel; Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: LJM716 — LJM716 (10-40 mg/kg) will be given as a once weekly infusion beginning on cycle 1 day 1. The doses of LJM716 will be increased as dose escalation proceeds until a maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) is established.
  Arms: LJM716-BYL719 arm
Drug: BYL719 — BYL719 (200-400 mg) will be administered orally on a once daily schedule starting cycle 1 day 1. The doses of BYL719 will be increased as dose escalation proceeds until a maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) is established.
  Arms: LJM716-BYL719 arm
Drug: Paclitaxel — In the Phase II portion of the study Paclitaxel is one of the 3 physician's choice drug which allows single-agent paclitaxel to be used per manufacturer's label.
  Arms: Paclitaxel, Docetaxel or Irinotecan arm
Drug: Docetaxel — In the Phase II portion of the study Docetaxel is one of the 3 physician's choice drug which allows single-agent docetaxel to be used per manufacturer's label.
  Arms: Paclitaxel, Docetaxel or Irinotecan arm
Drug: Irinotecan — In the Phase II portion of the study Irinotecan is one of the 3 physician's choice drug which allows single-agent irinotecan to be used per manufacturer's label
  Arms: Paclitaxel, Docetaxel or Irinotecan arm

SUMMARY:
To study the safety and efficacy of the combination of LJM716 and BYL719 against currently available treatments of physician's choice in previously treated esophageal squamous cell carcinoma patients.

DETAILED DESCRIPTION:
The study design included a Phase 1b dose escalation portion to define the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) for the combination of LJM716 and alpelisib, followed by an open-label, randomized Phase 2 part to compare anti-tumor activity of LJM716-alpelisib combination versus physician's choice of second-line therapy (paclitaxel, docetaxel, irinotecan). However, the phase 2 part was not conducted as the study was terminated early due to limited anti-tumor activity with LJM716-alpelisib combination observed in phase 1b.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma (ESCC)
* No more than one prior chemotherapy regimen for recurrent or metastatic ESCC (for Phase II only).
* Progression during or after platinum-based therapy for recurrent or metastatic ESCC, or recurrence within 6 months of platinum-based chemotherapy or chemoradiotherapy for localized disease.

Exclusion Criteria:

* Patients who received prior phosphoinositide-3-kinase (PI3K) inhibitor or anti-receptor tyrosine-protein kinase erbB-3 (ERBB3 or HER3) antibody treatment, including bi-specific antibodies with HER3 as one of the targets (patients with prior exposure to pertuzumab or epidermal growth factor receptor (EGFR)-targeted agents are eligible)
* Patients who do not have an archival or fresh tumor sample (or sections of it) available or readily obtainable.
* Patients with central nervous system (CNS) metastatic involvement.
* Patients who have received prior systemic anti-cancer treatment, such as cyclical chemotherapy or biological therapy within a period of time that is shorter than the cycle length used for that treatment (e.g. 6 weeks for nitrosourea, mitomycin-C) prior to starting study treatment.
* Patients who have received definitive radiotherapy ≤ 4 weeks prior to starting study drug, who have not recovered from side effects of such therapy and/or from whom ≥ 30% of the bone marrow was irradiated.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

PRIMARY OUTCOMES:
Phase Ib primary outcome measure: Incidence rate of dose limiting toxicities (DLTs). | approximately 8 months
  The open-label dose escalation part of the study will be guided by a well-established statistical method/model to estimate the maximum tolerated dose(s) and/or Recommended Phase II Dose (s) guided by the safety (incidence of dose limiting toxicities), efficacy, pharmacokinetics and pharmacodynamics data.
Phase II primary outcome measure: Progression free survival (PFS) | Every 6 weeks from the date of the baseline computed-tomography (CT) scan until the date of first documented evidence of disease progression or date of death, whichever comes first, assessed up to 24 months.
  Progression-free survival is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate assessment.

SECONDARY OUTCOMES:
Safety and tolerability of the LJM716-BYL719 | Every 21 days from the date of the baseline visit until the end of study visit (about 5 months)
  This will be assessed by looking at the number of Adverse Events (AEs), serious AEs (SAEs) changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions, reductions and dose intensity.
Best overall response (BOR), per RECIST 1.1 (Ph 1b ) | Every 21 days from the date of baseline computed tomography (CT) scan until end of treatment visit (about 4 months)
  BOR will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.
Plasma concentration versus time profiles Plasma PK parameters of LJM716, BYL719 | Baseline, 2hr,4hr,8hr,24hr,48hr,96hr, 168 hr, every 21 days for 10 cycles (21 days each) and at end of treatment (about 4 months)
  Plasma concentration versus time profiles Plasma PK parameters will be used to characterize the PK profiles of LJM716 and BYL719 when used in combination
Overall response rate (ORR) per RECIST 1.1 (Ph 1b ) | Every 21 days from the date of the baseline computed tomography (CT) scan until the end of treatment visit (about 4 months)
  Overall response rate will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.
Duration of response (DOR) per RECIST 1.1 (Ph 1b ) | Every 21 days from the date of the baseline computed tomography (CT) scan until the end of treatment visit (about 4 months)
  Duration of response will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.
Disease control rate (DCR) per RECIST 1.1 (Ph 1b ) | Every 21 days from the date of the baseline computed tomography (CT) scan until the end of treatment visit (about 4 months)
  Disease control rate will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.
Overall survival (OS) per RECIST 1.1 (for Ph 1b ) | Every 21 days from the date of the baseline computed tomography (CT) scan until the end of treatment visit (about 4 months)
  Overall survival will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.
Progression free survival (PFS) per RECIST 1.1 (Ph 1b ) | Every 21 days from the date of the baseline computed tomography (CT) scan until the end of study visit (about 5 months)
  Progression free survival will be used to further assess the anti-tumor activity of LJM716-BYL719 combination versus Paclitaxel, Docetaxel or Irinotecan.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (3):
  - University of Chicago Medical Center Dept of Onc, Chicago, Illinois
  - Karmanos Cancer Institute Dept of Onc, Detroit, Michigan
  - University of Texas/MD Anderson Cancer Center Gastrointestinal Med. Oncology, Houston, Texas
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLJM716X2103 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16294